CLINICAL TRIAL: NCT03467295
Title: Treatments and Outcomes of Untreated Cerebral Cavernous Malformations in CHINA (TOUCH): A Nationwide Multicenter Prospective Cohort Study.
Brief Title: Treatments and Outcomes of Untreated Cerebral Cavernous Malformations in CHina.
Acronym: TOUCH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Fuxin Lin, Principal Investigator, First Affiliated Hospital of Fujian Medical University
Other Study IDs: FAHFMU-2018-003
Record Dates: First submitted 2018-03-09; First posted 2018-03-16 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Cerebral Cavernous Malformations
Keywords: Cavernous Malformations, treatment.
MeSH Terms: conditions — Hemangioma, Cavernous, Central Nervous System | interventions — Surgical Procedures, Operative; Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgically treated group: Surgical removal of intracerebral CMs by craniotomy with or without following stereotactic radiosurgery.
  Interventions: Procedure: Surgery
- Conservatively treated group: Observation with the best medicine administration and supportive treatment are performed.
  Interventions: Procedure: Observation

INTERVENTIONS:
Procedure: Surgery — For patient in surgically treated group, surgical removal of intracerebral CMs by craniotomy is performed according to the principles as follows: less transgression of normal brain tissue; identification and protection of eloquent brain tissue; sparing associated developmental venous anomaly; hemosiderin rim resection for non-eloquent and superficial CMs and sparing yellowish tissue for eloquent and deep ones; Extended resections (mesial resection, standard temporal lobe resection) are recommend for epileptogenic CMs based on intra-operative EEG.
  Groups: Surgically treated group
Procedure: Observation — Observation is performed in conservatively treated patients with best medicine and supportive treatment, such as antiepileptic drugs, analgesic drugs and neurotrophic drugs. For patients with underlying diseases such as hypertension, hyperlipidemia or diabetes mellitus, after consulting with the relevant experts, the patients can be treated accordingly.
  Groups: Conservatively treated group

SUMMARY:
This nationwide multicenter prospective cohort study will collect the treatment information and outcomes of the patients with previously untreated cavernous malformations (U-CMs) in China (at least 2000 patients from 20 centers). The investigators aim to determine the effect of different treatments on long-term outcomes in patients with untreated cerebral cavernous malformations.

DETAILED DESCRIPTION:
Despite the availability of microsurgical excision and stereotactic radiosurgery for cavernoma treatment and known genetic causes of most familial forms of cavernoma, uncertainties remain about cause, diagnosis, prognosis, treatment, and care. According to the recently published CM treatment guideline, surgical and conservative treatments are both first-line therapeutic options in previously untreated CMs (U-CMs). However, given current data, neurosurgeons are still unable to counsel patients on which would be the best option. To address the absence of high level evidence to support cerebral CM treatment decisions, there is a need for a large sample size study of cerebral CM treatment with a prospective concurrent group. China has the largest population in the world and may have the most extensive and valuable clinical resources of U-CMs. But, till now, the current treatment and outcome situation of the disease in China is not well known. Thus, the investigators are conducting a nationwide multicenter prospective registry study in China to determine the effect of different treatments on long-term outcomes in patients with untreated cerebral cavernous malformations.At least 2000 patients with untreated cerebral cavernous malformation will be enrolled from 20 Grade Ⅲ A level hospitals distributed all over China. Clinical data and laboratory data are prospectively collected by electric case report form (CRF) and uploaded online by each neurosurgery center to form the prospective clinical database in First Affiliated Hospital of Fujian Medical University. This is a cohort follow-up study across a 5-year period with a 2 years interval of enrollment and 3 years follow up for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of cerebral CM on the basis of brain MRI or pathologic examination;
* Patients without any surgical intervention (microsurgery, radiosurgery, or multimodality treatment) before enrolment;
* Informed consent, and willing to accept long-term follow-up.

Exclusion Criteria:

* Patients receiving emergency surgery due to acute intracranial hematoma and resultant brain hernia;
* Patients with other never system diseases, such as aneurysms, tumors or other vascular malformations except venous development anomaly;
* Patients with severe underlying disease, which affects the patient's functional status and life expectancy;
* Patients with severe mental or psychologic disease.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with untreated cerebral cavernous malformation are enrolled from 20 Grade Ⅲ A level hospitals distributed all over China. At the time of the participants entered the study, lesions should not have been treated by surgery or radiosurgery previously. This is a cohort follow-up study across a 5-year period. All patients in this study should meet the inclusion and exclusion criteria. Informed written consent should be obtained from eligible adult patients or from the guardians of eligible pediatric patients. All patients in the prospective part of this study can withdraw at any time.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Poor outcome | 3 years
  The primary outcome of this study is patients with poor outcome (mRS>2 lasting at least 1year) at the last follow up.

SECONDARY OUTCOMES:
symptomatic hemorrhage | 3 years
  Requiring acute or subacute onset symptoms (any of headache, epileptic seizure, impaired consciousness, or new/worsened brain function deficit referable to the anatomic location of the CM) accompanied by radiological, pathological, surgical, or rarely only cerebrospinal fluid evidence of recent extra- or intralesional hemorrhage.
drug refractory epilepsy | 3 years
  Failure of adequate trials of two tolerated, appropriately chosen and used antiepileptic drug schedules (whether as monotherapies or in combination) to achieve sustained seizure freedom.
All-cause mortality | 3 years
  Death caused by all the causes

CONTACTS AND LOCATIONS:
Overall Officials: Dezhi Kang, MD,PHD, Study Chair — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The first affiliated hospital of fujian medical university, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
We will share individual participant data after the primary results have been published.

REFERENCES:
- [Derived] Li C, Huang S, Li Q, Zhuo L, Kang Y, Liu P, Huang W, Ma K, Lin X, Zhuang W, Chen D, Wang H, Yan L, Wang D, Lin Y, Kang D, Lin F. Plasma biomarkers in patients with familial cavernous malformation and their first-degree relatives: a cross-sectional study. Sci Rep. 2025 Apr 2;15(1):11284. doi: 10.1038/s41598-025-91141-6. PMID 40175401
- [Derived] Lin F, He Q, Gao Z, Yu L, Wang D, Zheng S, Lin Y, Kang D. Treatments and outcomes of untreated cerebral cavernous malformations in China: study protocol of a nationwide multicentre prospective cohort study. BMJ Open. 2020 Oct 29;10(10):e037957. doi: 10.1136/bmjopen-2020-037957. PMID 33122314